CLINICAL TRIAL: NCT06435325
Title: Effectiveness of a Precision Diet Based on Gene Expression Versus a Personalized Mediterranean-Style Diet in Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Principal Investigator, Jose Manuel Soria, Director of the Genomics Unit in Complex Diseases, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-SOB-2022-109
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-07

CONDITIONS: Overweight and Obesity
Keywords: Personalized nutrition; Epigenetics; Metabotype; Weight Loss; Well-being
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): The intervention arm will receive a hypocaloric Mediterranean-style diet (TEE - 500kcal, macronutrient distribution: 45 - 55% carbohydrates, 15 - 25% protein, and 25 - 35% fat) with dietary recommendations based on the participant's gene expression profile.
  Interventions: Behavioral: Precision diet
- Control arm (Active Comparator): The control arm will receive a hypocaloric Mediterranean-style diet (TEE - 500kcal, macronutrient distribution: 45 - 55% carbohydrates, 15 - 25% protein, and 25 - 35% fat) personalized to the participant's dietary and lifestyle habits.
  Interventions: Behavioral: Control diet

INTERVENTIONS:
Behavioral: Precision diet — After the recruitment and randomization, the participants will follow the assigned diet and recommendations for 3-months.
  Arms: Intervention arm
Behavioral: Control diet — After the recruitment and randomization, the participants will follow the assigned diet and recommendations for 3-months.
  Arms: Control arm

SUMMARY:
The present randomized controlled trial aims to evaluate the relationship between gene expression profiling and the response to a precision diet compared to a personalized Mediterranean-style diet (control diet) in metabolically healthy individuals with overweight and obesity.

Compared to the control diet, the precision diet is expected to increase adherence to dietary recommendations (resulting in weight loss and maintenance). In addition, the investigators postulate that the precision diet will lead to greater lifestyle changes, improving long-term well-being and health in people with overweight and obesity.

DETAILED DESCRIPTION:
The study aims to evaluate the effectiveness of a precision diet based on gene expression versus a personalized Mediterranean-style diet. For this purpose, a 12-week parallel randomized controlled trial will be conducted. Once eligible participants are recruited, each volunteer will attend two clinical visits (at baseline-week 0 [T0], and week 12 [T1]), a study initiation visit (at week 1), and three online follow-up visits (at weeks 3, 6 and 9).

First, the participants will come to the baseline visit [T0] in which, the investigators will collect data related to health status, body composition, lifestyle, and well-being. In addition, a registered nurse will collect a blood sample for gene expression profiling, along with other biochemical parameters, such as glycemic and lipid markers.

In the following days, the biochemical results from the baseline visit will be evaluated to confirm that the volunteers are metabolically healthy. For this reason, it will not be until seven days after the baseline visit that the eligibility of the participants will be confirmed. After this confirmation, participants will be scheduled for the study initiation visit.

At this visit, the volunteers will be randomly assigned to one of the two study arms, intervention (precision diet) or control diet. Those assigned to the intervention arm will follow the precision diet (a hypocaloric Mediterranean-style diet based on gene expression), while those assigned to the control arm will follow the control diet (a personalized hypocaloric Mediterranean-style diet without considering gene expression).

Then, 12 weeks after the start of the intervention, the end of the intervention [T1] will be scheduled, in which the investigators will evaluate the same variables as in the baseline visit [T0]. In addition, during the 12 weeks of the study, both groups will attend three online follow-up visits (every 3 weeks) to ensure adherence to the intervention, as well as continuous care and to adapt dietary recommendations when needed.

ELIGIBILITY:
Inclusion Criteria:

* BMI 26-35 Kg/m^2.
* Metabolically healthy.

Exclusion Criteria:

* Any comorbidity associated with obesity (such as type 2 diabetes mellitus, hypertension, dyslipidemia).
* Medications (Antidepressants; Antipsychotics; Anxiolytic; Statins; Antihypertensives; Insulin or anti-diabetics).
* Intragastric balloon or Bariatric surgery.
* History of weight loss treatment within the previous 3 months.
* Women with menopause, pregnancy, or breastfeeding.
* Smokers.
* Food allergies or intolerances.
* Eating disorders.
* Shift work.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in body mass index (BMI) from baseline to weeks 12. | Week 0 and 12.
  Calculated as weight (kg) divided by height (in squared meters), BMI= kg/m^2.
Changes in body fat from baseline to weeks 12. | Week 0 and 12.
  Measured as the percentage of body fat with a body composition analyzer (Inbody 120, Korea).

SECONDARY OUTCOMES:
Changes in gene expression profiling from baseline to weeks 12. | Week 0 and 12.
  The RNA from fasting blood samples will be sequenced using Illumina technology and then the Limma software package will be used to analyze gene expression data from the RNA sequence.
Changes in fasting blood lipids from baseline to weeks 12. | Week 0 and 12.
  Fasting measurement of triglycerides, total cholesterol, LDL-cholesterol and HDL-cholesterol (mmol/L) will be measured in venous blood with the standard methodology of the clinical analysis laboratory of the Hospital de Sant Pau.
Changes in glycemic markers from baseline to weeks 12. | Week 0 and 12.
  Fasting measurement of glucose, insulin, and glycated hemoglobin (mmol/L) will be measured in venous blood with the standard methodology of the clinical analysis laboratory of the Hospital de Sant Pau.
Changes in C-Reactive Protein (CRP) levels from baseline to weeks 12. | Week 0 and 12.
  Fasting measurement of CRP will be measured in venous blood with the standard methodology of the clinical analysis laboratory of the Hospital de Sant Pau.
Changes in waist and hip circumference from baseline to weeks 12. | Week 0 and 12.
  Measured to the nearest 0.1 cm using a flexible steel anthropometric tape (CESCORF, Brazil) calibrated in centimeters.
Changes in muscle mass from baseline to weeks 12. | Week 0 and 12.
  Measured as the kilograms of muscle mass with a body composition analyzer (Inbody 120, Korea).
Changes in physical activity from baseline to weeks 12. | Week 0 and 12.
  Measured in Metabolic Equivalents of Task (MET) per minute and week, using the short version of the International Physical Activity Questionnaire (IPAQ). The IPAQ consists of 7 questions that assess the frequency, duration, and intensity of physical activity (moderate and vigorous) performed in the last seven days, as well as walking and sitting time on a workday. The minimum value is 0 MET-minutes/week, indicating no physical activity. Higher scores represent a higher amount of physical activity, while lower scores indicate lower levels of physical activity.
Changes in energy and nutrient intake from baseline to week 12. | Week 0 and 12.
  Energy and nutrient intake will be assessed with a 151-item semi-quantitative food frequency questionnaire (FFQ) and a 3-day dietary record (DR), in which participants will record their food intake for three days. The frequency of consumption for each food item is reported on a nine-level incremental scale (never or almost never, 1-3 times per month, once per week, 2-4 times per week, 5-6 times per week, once per day, 2-3 times per day, 4-6 times per day and more than six times per day). To calculate energy and nutrient intake from both methods (FFQ and DR), the Spanish food composition tables will be used.
Changes in diet quality from baseline to week 12. | Week 0 and 12.
  Diet quality will be evaluated through the 17-item Mediterranean Diet Adherence Screener (MEDAS). The score ranges from 0 to 17, where higher scores indicate greater adherence to the Mediterranean Diet.
Changes in eating behavior from baseline to weeks 12. | Week 0 and 12.
  Eating behaviors will be measured with the Spanish version of the Three Factor Eating Questionnaire (TFEQ-R21). It consists of three subscales: Cognitive Restraint (CR), Uncontrolled Eating (UE), and Emotional Eating (EE). Scores range from 0 to 21 for CR and UE, and from 0 to 15 for EE. Higher scores on each subscale indicate higher levels of the corresponding eating behavior.
Changes in well-being from baseline to weeks 12. | Week 0 and 12.
  Well-being will be measured with the Spanish version of the World Health Organization (WHO-5) Well-being Index. Scores range from 0 to 25, where higher scores indicate higher well-being.
Changes in stress levels from baseline to week 12. | Week 0 and12.
  Stress will be evaluated through the Perceived Stress Scale (PSS-10), validated for Spanish population. Scores range from 0 to 40, where higher scores indicate a higher level of perceived stress.
Changes in depression and anxiety degree from baseline to week 12. | Week 0 and 12.
  Anxiety and depression state will be measured by the Hospital Anxiety and Depression Scale (HADS), validated for Spanish population. It consists of two subscales: HADS-A, designed to detect anxious states, and HADS-D, designed to detect depressive states. Scores range from o to 21, where higher scores indicate greater levels of anxiety or depression.
Changes in satiety from baseline to weeks 9. | Week 1 and 9.
  Satiety will be evaluated using the Visual Analogue Scale (VAS) after each meal. Scores range from 0 to 100 mm, where higher scores indicate greater levels of satiety.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Manuel Soria, Phd, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Maria Izquierdo-Pulido, Phd, Principal Investigator — University of Barcelona
Locations (1):
- Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain